CLINICAL TRIAL: NCT04721899
Title: Effect of Vitamin D on Vaginal / Endometrial Biomarkers and Endometrial Receptivity in Women With Fertility Problems
Brief Title: Vitamin D and Endometrial Receptivity in Infertile Women
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW19-134
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Infertility
Keywords: vitamin D; endometrial receptivity; infertility; recurrent pregnancy loss; recurrent implantation failure
MeSH Terms: conditions — Infertility | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vitamin D- recurrent implantation failure (RIF): All women will have endometrial biopsy twice- at baseline and after 8 weeks of taking vitamin D After 8 weeks of Vitamin D, a second endometrial biopsy using a Pipelle sampler will be collected from the patients 7 days after luteinizing hormone surge (LH+7) and the endometrial receptivity will be compared.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D- recurrent pregnancy loss (RPL): All women will have endometrial biopsy twice- at baseline and after 8 weeks of taking vitamin D After 8 weeks of Vitamin D, a second endometrial biopsy using a Pipelle sampler will be collected from the patients 7 days after luteinizing hormone surge (LH+7) and the endometrial receptivity will be compared.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D- infertility: All women will have endometrial biopsy twice- at baseline and after 8 weeks of taking vitamin D After 8 weeks of Vitamin D, a second endometrial biopsy using a Pipelle sampler will be collected from the patients 7 days after luteinizing hormone surge (LH+7) and the endometrial receptivity will be compared.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 50,000 IU once per week for 4 weeks, followed by 50,000 IU once every 2 weeks for 4 weeks

SUMMARY:
This is a prospective study comparing vaginal and endometrial biomarkers and the trophoblast spheroid attachment rate in women with fertility problems before and after taking Vitamin D for 8 weeks.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of vitamin D supplementation on vaginal / endometrial biomarkers and endometrial receptivity in women with fertility problems.

Women will have vaginal swab and endometrial biopsy twice. The first endometrial biopsy is performed using a Pipelle sampler 7 days after luteinizing hormone surge (LH+7) at baseline and the attachment rate of the trophoblast spheroid onto the isolated endometrial epithelial cells will be assessed to assess endometrial receptivity at baseline. Implantation biomarkers will be checked.

They will take Vitamin D 50,000 IU once per week for 4 weeks, followed by 50,000 IU once every 2 weeks for 4 weeks. After 8 weeks of Vitamin D, a second vaginal swab and endometrial biopsy using a Pipelle sampler by standard technique will be collected from the patients 7 days after luteinizing hormone surge (LH+7) and the endometrial receptivity will be compared.

The laboratory staff will not know whether the patient is taking any vitamin D when performing the trophoblast spheroid attachment assay/ biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age of women < 40years old
* Normal uterine cavity as demonstrated by pelvic scanning with or without saline infusion sonogram or hysteroscopy
* Regular ovulatory cycles

They will be divided into three groups:

* RIF patients (n=35)- those who have failed to get pregnant after replacing four or more cleavage stage embryos or two or more blastocysts in two consecutive transfers.
* RPL patients (n=35)- those who have failed in three pregnancies before 24 weeks of gestation and includes embryonic and fetal losses.
* 'Infertile group'(n=35)- infertility except RIF and RPL, e.g. those seeking for preimplantation genetic testing, male factor infertility, unexplained infertility.

Exclusion Criteria:

* History of any medical condition or medications that may predispose to vitamin D sensitivity, altered vitamin D metabolism and/ or hypercalcemia, including active tuberculosis or current therapy for tuberculosis, sarcoidosis, history of renal/ ureteral stones, parathyroid disease, renal or liver failure or current use of anti-convulsants
* Taking vitamin D supplement
* Endometrial polyp or fibroid distorting the uterine cavity
* Presence of hydrosalpinx not corrected surgically
* Refusal to join the study

  • Discontinuation criteria-
* If the woman becomes pregnant during the study
* Pelvic inflammatory disease/ uterine perforation after endometrial biopsy
* Vitamin D toxicity (hypercalcemia)
* Withdrawal by patient

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the Centre of Assisted Reproduction and Embryology, the University of Hong Kong at Queen Mary Hospital. Infertile women who are in the waiting list for IVF or have failed one IVF cycle will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in endometrial receptivity | 8 weeks
  Assessed by the attachment rate of trophoblast spheroid attachment assay onto the isolated endometrial epithelial cells

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided